CLINICAL TRIAL: NCT02244827
Title: A Phase I, Open Label, Single Dose Study to Evaluate The Pharmacokinetics of WCK 2349 In Patients With Hepatic Impairment
Brief Title: Pharmacokinetics of WCK 2349 In Patients With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: W-2349-102
Record Dates: First submitted 2014-09-10; First posted 2014-09-19 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — levonadifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WCK 2349 (Experimental): Each subject will receive a single oral dose of WCK 2349 1000 mg (i.e., 2 tablets of 400 mg and 1 tablet of 200 mg) with 240 mL water on Day 1 in the morning. Study drug will be administered after a fast of at least 8 hours.
  Interventions: Drug: WCK 2349

INTERVENTIONS:
Drug: WCK 2349 — levonadifloxacin (active drug) and the sulfate metabolite
  Other Names: levonadifloxacin (active drug)

SUMMARY:
This study is aimed to compare the pharmacokinetics of levonadifloxacin and its sulfate metabolite after a single dose of oral WCK 2349 1000 mg in patients with hepatic impairment and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI): 18.0 - 38.0 (Body weight in kg / Height in m2), both inclusive.
* Subjects must fulfill the following criteria:

Patients with hepatic impairment:

* Considered clinically stable in the opinion of the Investigator
* Patients with different degrees of impaired hepatic function as assessed by a Child-Pugh classification score: mild (5-6 points), moderate (7-9 points) and severe (10-15 points) impaired hepatic function.
* Documented history of cirrhosis diagnosed by liver biopsy, ultrasonography (USG), computed tomography (CT) scan, or magnetic resonance imaging (MRI) OR

Healthy volunteers:

* Have normal hepatic function
* Participants with a history of self-limited hepatitis A with complete resolution documented at least 6 months prior to entry will be allowed

Exclusion Criteria:

* Known hypersensitivity to quinolones/fluoroquinolones.
* Subjects must not fulfill the following criteria:

In hepatically impaired patients:

* Use of prohibited concomitant medication, with the exception of those essential for the management of hepatic impairment and the treatment of concomitant stable medical conditions for the hepatically impaired patients as per the discretion of the Investigator.
* Fluctuating or rapidly deteriorating hepatic function as indicated by recent history or widely varying or worsening of clinical and/or laboratory signs of hepatic impairment as judged by the Investigator.
* Concomitant treatment with Interferon or other prohibited medications
* Active stage 3 and stage 4 encephalopathy OR

Healthy Volunteers:

* Use of any concomitant medication within 7 days from the screening except those deemed safe for the study by the Investigator and Medical Monitor.
* History of any clinically significant chronic and/or active hepatic disease including elevations of serum transaminases including aspartate aminotransferase (AST) and alanine aminotransferase (ALT) [except those which are considered non-significant by the Investigator; however, these should not exceed 1.5 times the Upper Limit of Normal (ULN)], hepatitis (Hepatitis A, B or C), biliary tract disease, or history of any significant gastrointestinal surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To compare the pharmacokinetics parameters -AUC,Cmax, tmax, λz, t1/2, systemic clearance and apparent volume of distribution. | 48 hours
  To compare the pharmacokinetics of levonadifloxacin and its sulfate metabolite after a single dose of oral WCK 2349 in patients with hepatic impairment and healthy volunteers

SECONDARY OUTCOMES:
To evaluate the safety and tolerability parameters- Number of AE , Vital signs, clinical laboratory values, abnormal physical examinations and ECGs | 7 weeks
  To evaluate the safety and tolerability of oral WCK 2349 in patients with hepatic impairment and healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Preston, M.D., Principal Investigator — Division of Clinical Pharmacology,University of Miami
Locations (1):
- University of Miami,Division of Clinical Pharmacology, Miami, Florida, United States